CLINICAL TRIAL: NCT04961580
Title: Pharmacokinetics and Pharmacodynamics of Ceftazidime Avitbatan Sodium in Children With Severe Infection
Brief Title: PK/PD of Ceftazidime Avitbatan Sodium in Children With Severe Infection
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-23
Record Dates: First submitted 2021-07-05; First posted 2021-07-14 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Sepsis; Antibiotic Reaction
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ceftazidime avitbatan sodiumt group: Children treated with ceftazidime avitbatan sodium in the pediatric intensive care unit will be enrolled in this group. Blood sample will be retained at various time intervals for pharmacokinetics.
  Interventions: Drug: Ceftazidime Avitbatan Sodium

INTERVENTIONS:
Drug: Ceftazidime Avitbatan Sodium — For 6-18 years children, 62.5 mg/kg/once，q8h ; 3-6 months of age 50 mg/kg/ once,q8h, intravenous administration for 2 hours, daily dose is not more than 2.5g, children will be administrated at least five times.

SUMMARY:
Ceftazidime avitbatan sodium is a broad-spectrum antibiotic with an antimicrobial spectrum covering resistant gram-negative bacteria. Its use in pediatric intensive care for severe infections is not unusual. Pathophysiological changes in severe sepsis can lead to significant changes in pharmacokinetics and pharmacodynamics during continuous renal replacement therapy.This research aims to study change of pharmacokinetic and pharmacodynamic in severe infection children with extracorporeal life support, thus improve the treatment of severe sepsis and sepsis shock.

DETAILED DESCRIPTION:
This study is an observational clinical study. Subjects were recruited from children with severe infection receiving ceftazidime avitbatan sodium under routine clinical diagnosis and treatment routine. There is no control, no double-blind randomized design, and the normal treatment schedule of patients was not interfered with, and the disease risk of patients was not increased.All subjects had received at least 5 doses of ceftazidime avitbatan Sodium before enrollment.

Blood sampling time points of ceftazidime avitbatan sodium are listed as follow:

Before administration (0 min); 5,30 min,1 h,2 h,4 h and 8 h after administration, if blood purification is received, one blood sample will be collected before and after the filter at the same time point.

The concentration of ceftazidime avitbatan sodium in whole blood will be analyzed at Huashan Hospital of Fudan University.

ELIGIBILITY:
Inclusion Criteria:

* Children who are admitted in the pediatric intensive care unit receiving ceftazidime avitbatan sodium

Exclusion Criteria:

* No Informed Consent signed
* Participate in other clinical trials

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children receiving cefatadine and averbactam sodium in pediatric intensive care unit including but not limited to children with liver insufficiency, hypoproteinemia, ECMO treatment, CRRT treatment or sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) Pharmacokinetic Parameter | Day 1-5
  Time to reach the maximum plasma concentration (Tmax) after administrations of a single dose and multiple doses of the study drug

SECONDARY OUTCOMES:
Terminal Phase Elimination Half-life (T1/2) Pharmacokinetic Parameter | Day 1-5
  Time required for half of the drug to be eliminated from the plasma after administration of a single dose of the study drug.
AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity Pharmacokinetic Parameter | Day 1-5
  Area under the plasma concentration-time curve from time 0 to infinity after administration of a single dose of the study drug
AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Pharmacokinetic Parameter | Day1-5
  Area under the curve from 0 to 24 hours after administrations of a single dose and multiple doses of the study drug
Cmax: Maximum Observed Plasma Concentration Pharmacokinetic Parameter | Day1-5
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration after administrations of a single dose and multiple doses of the study drug

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Lu, doctor, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's hosptial of fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No